CLINICAL TRIAL: NCT06789432
Title: Efficacy and Safety of Atorvastatin and Ezetimibe (10/10mg) Fixed Dose Combination Versus Atorvastatin (20mg) Monotherapy in Bangladeshi Population
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Md. Alimur Reza (Industry)
Responsible Party: Sponsor-Investigator, Dr. Md. Alimur Reza, Epidemiologist, Beximco Pharmaceuticals Ltd.
Organization: Beximco Pharmaceuticals Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEX2411001
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hyperlipidemia (E.G., Hypercholesterolemia)
Keywords: increased LDL-C level; Hyperlipidemia; Atorvastatin (10 mg) and Ezetimibe (10 mg)
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-centred, open-label, randomized controlled trial in patients with increased LDL-C levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Atorvastatin 10 mg and ezetimibe 10 mg
- Arm 2 (Experimental)
  Interventions: Drug: Atorvastatin 20 mg

INTERVENTIONS:
Drug: Atorvastatin 10 mg and ezetimibe 10 mg — Atorvastatin/Ezetimibe 10/10mg once daily
  Arms: Arm 1
Drug: Atorvastatin 20 mg — Atorvastatin (20 mg) Monotherapy once daily
  Arms: Arm 2

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of a fixed-dose combination of atorvastatin (10 mg) and ezetimibe (10 mg) compared to atorvastatin (20 mg) monotherapy in the Bangladeshi population.

Researchers will compare atorvastatin (10 mg) and ezetimibe (10 mg) to atorvastatin (20 mg) monotherapy to see if atorvastatin (10 mg) and ezetimibe (10 mg) FDC works to treat dyslipidemia.

Participants will:

* Take a fixed-dose combination of atorvastatin (10 mg) and ezetimibe (10 mg) compared to atorvastatin (20 mg) monotherapy for 3 months
* Follow-up visits at 6 weeks and 12 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years.
* Patients with a confirmed diagnosis of elevated LDL-C levels necessitating medical management.
* Patients in the low to moderate cardiovascular disease (CVD) risk category according to ESC guidelines (2019)

  * Low-risk: Increased LDL-C level without any co-morbidities
  * Moderate-risk: Young patients (T1DM <35 years; T2DM <50 years) with DM duration <10 years, without other risk factors.

Exclusion Criteria:

* History of hypersensitivity to any study drugs.
* Clinically significant hepatic impairment (ALT, AST level > 2xULN) and/or renal impairment (Serum creatinine level ≥2xULN).
* Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) with cirrhosis, end-stage liver disease, cancer, psychiatric instability, HIV + status, intestinal malabsorption.
* Pregnant or lactating females.
* The presence of a condition that, in the opinion of the investigator, would place the subject at increased risk from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in LDL-C from baseline | Baseline to Week 12
  Compare the mean change in LDL-C (mg/dL) from baseline to week 12 in both groups.
Percentage of patients withdrawn from the study | Baseline to Week 12
  Compare the percentage of patients withdrawn from the study due to adverse events in two groups.

SECONDARY OUTCOMES:
Achievement of target levels of LDL-C | Baseline to Week 12
  Compare the frequency of achieving the target levels of LDL-C in both groups after 12 weeks
Mean changes in total cholesterol (TC), HDL-C and TG | Baseline to Week 12
  Compare the mean changes in total cholesterol (TC), HDL-C and TG from baseline to week 12 in both arms.
Frequency of myopathy | Baseline to Week 12
  Compare the frequency of myopathy after 12 weeks between two arms
Frequency of AEs & SAEs | Baseline to Week 12
  Compare the frequency of AEs & SAEs between two arms
Changes in SGPT Levels in Both Arms | Baseline to Week 12
  Compare the change in SGPT (U/L) levels in both arms.
Changes in Serum Creatinine Levels in Both Arms | Baseline to Week 12
  Compare the changes in SGPT (U/L) levels in both arms.
Changes in creatine phosphokinase (CPK) level in Both Arms | Baseline to Week 12
  Compare the changes in creatine phosphokinase (CPK) level in Both Arms

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Abdullah Al Shafi Majumder, MD, FACC, FRCP (E), FRCP (G), Principal Investigator — Professor, Dept. of Cardiology, Popular Medical College, Dhaka.
Locations (1):
- Popular Medical College & Hospital, Dhaka, Dhaka Division, Bangladesh